CLINICAL TRIAL: NCT04272242
Title: Drug-Drug Interactions Between Rifapentine and Dolutegravir in HIV/LTBI Co-Infected Individuals
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Opening of Arm 2 was dependent upon assessment of DTG pharmacokinetics (PK) data from participants in Arm 1. Arm 1 is complete and results are reported. Arm 2 was not conducted based on the Arm 1 PK assessment.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5372; 38485 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: HIV Infection; LTBI
Keywords: LTBI; HIV and LTBI Co-Infection; Rifapentine; Dolutegravir Interaction
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir; Isoniazid; rifapentine; Antiretroviral Therapy, Highly Active; Pyridoxine; Vitamin B 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: DTG + INH + RPT (Experimental): Participants received 50 mg of DTG orally twice daily (~12 hours apart). Participants received 300 mg of INH and 600 mg of RPT orally each morning for 4 weeks.
  Participants also received 25 or 50 mg of pyridoxine (vitamin B6) with each dose of INH.
  Participants remained on DTG-based ARV treatment with 2 NRTIs (excluding TAF) during the study. Participants took non-study supply of DTG for morning doses, and study-supplied DTG for evening doses.
  Interventions: Drug: Dolutegravir (DTG); Drug: Isoniazid (INH); Drug: Rifapentine (RPT); Drug: Antiretroviral Therapy (ART); Dietary Supplement: Pyridoxine (Vitamin B6)
- Arm 2: DTG + INH + RPT (Experimental): Participants were to receive 50 mg of DTG orally each morning and 300 mg of INH and 600 mg of RPT orally each morning for 4 weeks.
  Participants were also to have received 25 or 50 mg of pyridoxine (vitamin B6) with each dose of INH.
  Participants were to remain on once-daily DTG-based ARV treatment with 2 NRTIs (excluding TAF) during the study with DTG supplied from non-study ARV supply.
  It was decided to not move forward with Arm 2 of the study based on the Arm 1 PK assessment and no participants were enrolled in Arm 2.
  Interventions: Drug: Dolutegravir (DTG); Drug: Isoniazid (INH); Drug: Rifapentine (RPT); Drug: Antiretroviral Therapy (ART); Dietary Supplement: Pyridoxine (Vitamin B6)

INTERVENTIONS:
Drug: Dolutegravir (DTG) — Administered orally
Drug: Isoniazid (INH) — Administered orally
Drug: Rifapentine (RPT) — Administered orally
Drug: Antiretroviral Therapy (ART) — Participants remained on DTG-based ARV treatment with 2 NRTIs (excluding TAF) during the study. NRTIs were not provided by the study. Arm 1 participants took non-study supply of DTG for morning doses, and study-supplied DTG for evening doses. For Arm 2 participants, DTG was to have come from non-study ARV supply.
Dietary Supplement: Pyridoxine (Vitamin B6) — Participants received 25 or 50 mg of pyridoxine (vitamin B6) with each dose of INH, based on the current local, national, or international dosing guidelines. Pyridoxine was not provided by the study.

SUMMARY:
This study evaluated the potential drug-drug interactions between dolutegravir (DTG) and steady state rifapentine (RPT) when RPT was given with isoniazid (INH) daily for 4 weeks (1HP) as part of treatment for latent TB infection (LTBI) in HIV-1 and LTBI co-infected individuals.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the potential drug-drug interactions between dolutegravir (DTG) and steady state rifapentine (RPT) when RPT was given with isoniazid (INH) daily for 4 weeks (1HP) as part of treatment for latent TB infection (LTBI) in HIV-1 and LTBI co-infected individuals.

Participants received study-provided INH and RPT once daily for 4 weeks (1HP). During the 1HP treatment, DTG was administered twice daily in Arm 1. Arm 2 planned to administer DTG once daily.

At study entry, all participants were required to be on DTG-based antiretroviral (ARV) treatment with 2 nucleoside reverse transcriptase inhibitors (NRTIs) (tenofovir alafenamide [TAF] was prohibited) during the study. In Arm 1, DTG 50 mg was administered twice daily; the morning dose from non-study ARV supply and the evening dose from study supply.

Participants were also required to receive pyridoxine (vitamin B6) with each dose of INH based on the current local, national, or international dosing guidelines. NRTI therapy and pyridoxine (vitamin B6) was not provided by the study.

The majority of Arm 1 participants were on study for 6 weeks (a 4-week on-study treatment period and a 2-week follow-up period). Arm 1 participants could be on study for up to 11 weeks if the on-study treatment duration was extended or if participants needed additional follow-up visits to measure viral load.

The study began enrollment with Arm 1. Opening of Arm 2 was dependent upon assessment of DTG pharmacokinetics (PK) data from participants in Arm 1.

Arm 1 is complete and results are reported. Arm 2 was not conducted based on the Arm 1 PK assessment.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness of participant or legal guardian/representative to provide informed consent.
* Weight ≥40 kg and a body mass index (BMI) of greater than 18.5 kg/m^2.
* Documentation of HIV-1 infection status, as below:

  * HIV-1 infection, documented by any licensed rapid HIV test or HIV-1 E/CIA test kit at any time prior to entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen or plasma HIV-1 RNA viral load. Two or more HIV-1 RNA viral loads of >1,000 copies/mL are also acceptable as documentation of HIV-1 infection.
  * Note A: The term "licensed" refers to a US Food and Drug Administration (FDA)-approved kit, which is required for all investigational new drug (IND) studies, or for sites that are located in countries other than the United States, a kit that has been certified or licensed by an oversight body within that country and validated internally. Non-US sites are encouraged to use US FDA-approved methods for IND studies.
  * Note B: World Health Organization (WHO) and Centers for Disease Control and Prevention (CDC) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.
* HIV-1 plasma viral load <50 copies/mL obtained within 30 days prior to study entry by any US laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent, or at any network-approved non-US laboratory that is Virology Quality Assessment (VQA) certified.
* At US sites: Evidence of LTBI by tuberculin skin test (TST) reactivity ≥5 mm, or a positive interferon gamma release assay (IGRA) at any time prior to study entry.

  * At non-US sites: Indication for LTBI treatment according to WHO latent TB guidelines (Note: TST/IGRA results not required).
* On a stable once daily DTG (50 mg) based ART with once daily 2 NRTIs and

  * with at least 28 total days of DTG and NRTI dosing prior to study entry
  * with no gaps in self-reported DTG and NRTI adherence of more than 3 consecutive days in the 28 days prior to study entry
  * with no intention to change ART for the duration of the study
  * NOTE A: Participants who switch from another ART regimen to DTG to meet eligibility requirements for this study will be eligible to enroll as long as the ART is switched at least 28 days prior to study entry.
* Chest radiograph or chest computed tomography (CT) scan performed within 30 days prior to study entry without evidence of active TB.

  * NOTE: An existing chest X-ray or CT scan from within 30 days prior to entry can be used as qualifying chest imaging. If chest imaging will be performed for study evaluation (i.e., Screening), then chest X-ray should be performed. A CT scan will be used only if an existing scan is already available and will not be performed as part of study.
* The following laboratory values obtained within 30 days prior to study entry by any US laboratory that has a CLIA certification or its equivalent, or at any network approved non-US laboratory that operates in accordance with Good Clinical Laboratory Practice (GCLP) and participates in appropriate external quality assurance programs.

  * Absolute neutrophil count (ANC) >750 cells/mm^3
  * Hemoglobin ≥7.4 g/dL
  * Platelet count ≥50,000/mm^3
  * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) <2.5 X the upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) <2.5 X ULN
  * Total bilirubin ≤1.5 x ULN
  * Creatinine <1.3× ULN
* For females of reproductive potential, negative serum or urine pregnancy test at Screening within 30 days prior to entry and within 48 hours prior to entry by any US clinic or laboratory that has a CLIA certification or its equivalent, or is using a point of care (POC)/CLIA-waived test, or at any network-approved non-US laboratory or clinic that operates in accordance with GCLP and participates in appropriate external quality assurance programs.

  * NOTE A: If screening visit occurs within 48 hours prior to entry, only one test will occur prior to entry.
  * NOTE B: Urine test must have a sensitivity of 15-25 mIU/mL.
* Female participants of reproductive potential must agree not to participate in the conception process (i.e., active attempt to become pregnant, in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, must agree to use one reliable nonhormonal method of contraception, as listed below, while on study treatment and through study completion.
* Acceptable forms of contraception include:

  * Intrauterine device (IUD) or intrauterine system
  * Cervical cap with spermicide
  * Diaphragm with spermicide
  * Condoms (male or female)
  * NOTE A: Hormonal methods may be used, however, one of the other acceptable forms of contraception listed above must also be used through the duration of the study because of potential interactions with RPT.
  * NOTE B: Participant-reported history is acceptable documentation of menopause (i.e., at least 1 year amenorrheic), hysterectomy, or bilateral oophorectomy or bilateral tubal ligation; these candidates are considered not of reproductive potential and are eligible without the required use of contraception.

Exclusion Criteria:

* Breastfeeding, pregnancy, or plans to become pregnant.
* Known allergy/sensitivity or any hypersensitivity to components of the study drugs, or their formulations.
* Presence of any confirmed or probable active TB based on criteria listed in the current AIDS Clinical Trials Group (ACTG) Diagnosis Appendix at screening.
* History of rifamycin-monoresistant, INH-monoresistant, multi-drug resistant (MDR) or extensively-drug resistant (XDR) TB at any time prior to study entry
* Known exposure to rifamycin-monoresistant, INH-monoresistant, MDR- or XDR-TB (e.g., household member of a person with rifamycin-monoresistant, INH monoresistant, MDR- or XDR-TB) at any time prior to study entry by participant self report or medical records.
* History of peripheral neuropathy Grade ≥2 according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, July 2017, which can be found on the DAIDS RSC website at https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Acute or serious illness requiring systemic treatment and/or hospitalization within 7 days prior to study entry.
* Known cirrhosis, a history of decompensated liver disease (ascites, hepatic encephalopathy, or esophageal varices) or current Child Pugh Class B or C hepatic impairment.

  * Note: Refer to the study protocol for Child Pugh scoring and classification table.
* Initiated, discontinued, or changed doses of drugs that are P-glycoprotein (PGP) inducers, that are P-glycoprotein (PGP) inhibitors,or that are known to have drug interactions with DTG, within 30 days prior to study entry.

  * Note: Refer to the list of prohibited and precautionary medications in the study protocol.
* Known porphyria at any time prior to study entry.
* Receipt of any other antiretroviral therapy other than DTG and 2 NRTI within 28 days prior to study entry.
* Receipt of TAF within 28 days prior to study entry.
* Documented resistance that may confer reduced susceptibility to DTG, at any time prior to study entry. This includes the following INSTI mutations: Q148 substitutions, T66A, L74I/M, E138A/K/T, G140S/A/C, Y143R/C/H, E157Q, G163S/E/K/Q, G193E/R, or N155H.
* Clinically suspected INSTI resistance, at any time prior to study entry, as evidenced by prior receipt of INSTI containing ART, during which time two or more HIV-1 RNA levels of >200 copies/mL were observed after having attained virologic suppression to <200 copies/mL and without known interruption.
* Consumption of >3 alcohol beverages on any day within 30 days prior to entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-02-27 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Podany, PharmD, Study Chair — University of Nebraska
Locations (10):
- United States (2):
  - University of California HIV/AIDS CRS, San Francisco, California
  - Houston AIDS Research Team CRS, Houston, Texas
- Gaborone CRS, Gaborone, South-East District, Botswana
- Haiti (2):
  - GHESKIO Institute of Infectious Diseases and Reproductive Health (GHESKIO - IMIS) CRS, Port-au-Prince
  - Les Centres GHESKIO Clinical Research Site (GHESKIO-INLR) CRS, Port-au-Prince
- Malawi CRS, Lilongwe, Central Malawi, Malawi
- South Africa (2):
  - University of Cape Town Lung Institute (UCTLI) CRS, Cape Town
  - South African Tuberculosis Vaccine Initiative (SATVI) CRS, Cape Town
- Thai Red Cross AIDS Research Centre (TRC-ARC) CRS, Pathum Wan, Bangkok, Thailand
- Milton Park CRS, Milton Park, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://submit.mis.s-3.net/ Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.

REFERENCES:
- [Derived] Podany AT, Cramer Y, Imperial M, Rosenkranz SL, Avihingsanon A, Arduino R, Samaneka W, Gelmanova I, Savic R, Swindells S, Dawson R, Luetkemeyer AF. Twice-Daily Dolutegravir-Based Antiretroviral Therapy With 1 Month of Daily Rifapentine and Isoniazid for Tuberculosis Prevention. Clin Infect Dis. 2024 Oct 15;79(4):983-989. doi: 10.1093/cid/ciae183. PMID 38568956
- See also: Location of Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017 — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in Arm 1 were enrolled from February 2021 to November 2021 at 9 selected US and non-US ACTG clinical research sites. It was decided to not move forward with Arm 2 of the study and no participants were enrolled in Arm 2. Results are for Arm 1 only.
Pre-assignment Details: Participants were not randomized and enrollment was not stratified. To create by-country diversity of participants, screening and accrual limits were set for US and non-US sites.
Groups:
- Arm 1: DTG + INH + RPT: Participants received 50 mg of DTG orally twice daily (~12 hours apart). Participants received 300 mg of INH and 600 mg of RPT orally each morning for 4 weeks.
  Participants also received 25 or 50 mg of pyridoxine (vitamin B6) with each dose of INH.
  Participants remained on DTG-based ARV treatment with 2 NRTIs (excluding TAF) during the study. Participants took non-study supply of DTG for morning doses, and study-supplied DTG for evening doses.
  Dolutegravir (DTG): Administered orally
  Isoniazid (INH): Administered orally
  Rifapentine (RPT): Administered orally
  Antiretroviral Therapy (ART): Participants remained on DTG-based ARV treatment with 2 NRTIs (excluding TAF) during the study. NRTIs were not provided by the study. Arm 1 participants took non-study supply of DTG for morning doses, and study-supplied DTG for evening doses. For Arm 2 participants, DTG was to have come from non-study ARV supply.
  Pyridoxine (Vitamin B6): Participants received 25 or 50 mg of pyridoxine (vitamin B6) with each dose of INH, based on the current local, national, or international dosing guidelines. Pyridoxine was not provided by the study.
Period: Overall Study
Arm/Group | Arm 1: DTG + INH + RPT
Started | 37
Completed | 32
Not Completed | 5
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All participants who enrolled to the study
Arm/Group | Arm 1: DTG + INH + RPT
Number analyzed (Participants) | 37
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41.0 [35.0 to 48.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 25
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Haiti | 3
  United States | 4
  Malawi | 4
  Botswana | 3
  South Africa | 7
  Zimbabwe | 8
  Thailand | 8
HIV-1 RNA below 50 copies/mL [Count of Participants; unit: Participants]
  Below 50 copies/mL | 36
  50 copies/mL or Greater | 1

OUTCOME MEASURES:

1. Primary Outcome: DTG PK Parameter Maximum Plasma Concentration (Cmax) Determined Based on DTG Levels From Individual Participants in Arm 1 by Visit Day
Description: This evaluates the effect of RPT on the DTG PK parameter Cmax obtained from participants enrolled in Arm 1 at day 0 (DTG QD) and day 28 (DTG BID with 1HP). Cmax defines the model-predicted maximum concentration observed over the 12- or 24- hours of the DTG dosing interval.
Time Frame: Intensive DTG PK samples at pre-dose, 1h, 2h, 4h, 8h, 12h, 13h, 14h, 23h and 24h post-dose at days 0 and 28
Population: All Arm 1 participants who initiated the 1HP TB regimen, who completed 28 daily doses RPT/INH within the 6-week study period, and who took DTG twice-daily for days 1-28. Sampling took place after ensuring 3 days of consecutive DTG QD dosing prior to day 0, and 3 days of consecutive DTG BID with 1HP dosing prior to Day 28.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm 1: DTG + INH + RPT
Number analyzed (Participants) | 32
ng/mL
  Day 0 | 4180.8 [3920.6 to 5196.4]
  Day 28 | 3913.5 [3475.7 to 4743.1]
Statistical Analysis 1: Comparison: Arm 1: DTG + INH + RPT; Statistical analysis for Cmax, comparing Day 28 to Day 0; Test type: Equivalence — GMRs and associated 90% confidence intervals were calculated to assess the overall effect of 1HP on DTG PK; Geometric Mean Ratio = 0.92, 90% CI 2-sided [0.91 to 0.93] — The numerator represents Day 28 and the denominator represents Entry

2. Primary Outcome: DTG PK Parameter Area Under the Concentration Time Curve (AUC0-24) Calculated Based on Intensive PK Samples Obtained From Individual Participants Enrolled in Arm 1 by Visit Day
Description: This evaluates the effect of RPT on the DTG PK parameter AUC 0-24h obtained from participants enrolled in Arm 1 at day 0 (DTG QD) and day 28 (DTG BID with 1HP). AUC 0-24h defines area under the concentration-time curve over the period of 24 hours post-dose estimated based on the fitted model. For Arm 1, Day 28 (BID dosing), participant-specific AUC0-24h was estimated by summing participant-specific estimated AUC values for the 0-12 hour dosing interval (AUC0-12).
Time Frame: Intensive DTG PK samples at pre-dose, 1h, 2h, 4h, 8h, 12h, 13h, 14h, 23h and 24h post-dose at days 0 and 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: h*ng/mL
Arm/Group | Arm 1: DTG + INH + RPT
Number analyzed (Participants) | 32
h*ng/mL
  Day 0 | 68079.5 [59139.5 to 85561.0]
  Day 28 | 65261.3 [56748.6 to 81999.4]
Statistical Analysis 1: Comparison: Arm 1: DTG + INH + RPT; Statistical analysis for AUC0-24, comparing Day 28 to Day 0; Test type: Equivalence — GMRs and associated 90% confidence intervals were calculated to assess the overall effect of 1HP on DTG PK; Geometric Mean Ratio = 0.96, 90% CI 2-sided [0.96 to 0.96] — The numerator represents Day 28 and the denominator represents Entry

3. Primary Outcome: DTG PK Parameter Minimum Plasma Concentration (Cmin) Determined Based on DTG Levels From Individual Participants in Arm 1 by Visit Day
Description: This evaluates the effect of RPT on the DTG PK parameter Cmin obtained from participants enrolled in Arm 1 at day 0 (DTG QD) and day 28 (DTG BID with 1HP). Cmin defines the model-predicted minimum concentration observed over the 12- or 24- hour DTG dosing interval.
Time Frame: Intensive DTG PK samples at pre-dose, 1h, 2h, 4h, 8h, 12h, 13h, 14h, 23h and 24h post-dose at days 0 and 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm 1: DTG + INH + RPT
Number analyzed (Participants) | 32
ng/mL
  Day 0 | 1726.1 [1267.9 to 2395.6]
  Day 28 | 1717.5 [1206.6 to 2502.7]
Statistical Analysis 1: Comparison: Arm 1: DTG + INH + RPT; Statistical analysis for Cmin, comparing Day 28 to Day 0; Test type: Equivalence — GMRs and associated 90% confidence intervals were calculated to assess the overall effect of 1HP on DTG PK; Geometric Mean Ratio = 0.99, 90% CI 2-sided [0.97 to 1.00] — The numerator represents Day 28 and the denominator represents Entry

4. Primary Outcome: DTG PK Parameter Ctrough Determined Based on DTG Levels From Individual Participants in Arm 1 at Day 28
Description: This evaluates the effect of RPT on the DTG PK parameter Ctrough obtained from participants enrolled in Arm 1 at day 28 (DTG BID with 1HP). Ctrough defines the observed non-model based minimum concentration observed over the 12- hour DTG dosing interval.
Time Frame: Intensive DTG PK samples at pre-dose, 1h, 2h, 4h, 8h, 12h, 13h, 14h, 23h and 24h post-dose at day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Arm 1: DTG + INH + RPT
Number analyzed (Participants) | 32
ng/mL | 1987.0 [1331.0 to 2377.5]

5. Primary Outcome: DTG PK Parameter Maximum Plasma Concentration (Cmax) Determined Based on DTG Levels From Individual Participants in Arm 2 by Visit Day
Description: This evaluates the effect of RPT on the DTG PK parameter Cmax obtained from participants enrolled in Arm 2 at day 0 (DTG QD) and day 28 (DTG QD with 1HP). Cmax defines the model-predicted maximum concentration observed over the 24- hours of the DTG dosing interval.
Time Frame: Intensive DTG PK samples at pre-dose, 1h, 2h, 4h, 8h, 12h, 23h and 24h post-dose at days 0 and 28
Population: It was decided to not move forward with Arm 2 of the study and no participants were enrolled in Arm 2.
Groups:
- Arm 2: DTG + INH + RPT: Participants were to receive 50 mg of DTG orally each morning and 300 mg of INH and 600 mg of RPT orally each morning for 4 weeks.
  Participants were also to have received 25 or 50 mg of pyridoxine (vitamin B6) with each dose of INH.
  Participants were to remain on once-daily DTG-based ARV treatment with 2 NRTIs (excluding TAF) during the study with DTG supplied from non-study ARV supply.
  It was decided to not move forward with Arm 2 of the study based on the Arm 1 PK assessment and no participants were enrolled in Arm 2.
  Dolutegravir (DTG): Administered orally
  Isoniazid (INH): Administered orally
  Rifapentine (RPT): Administered orally
  Antiretroviral Therapy (ART): Participants remained on DTG-based ARV treatment with 2 NRTIs (excluding TAF) during the study. NRTIs were not provided by the study. Arm 1 participants took non-study supply of DTG for morning doses, and study-supplied DTG for evening doses. For Arm 2 participants, DTG was to have come from non-study ARV supply.
  Pyridoxine (Vitamin B6): Participants received 25 or 50 mg of pyridoxine (vitamin B6) with each dose of INH, based on the current local, national, or international dosing guidelines. Pyridoxine was not provided by the study.
Arm/Group | Arm 2: DTG + INH + RPT
Number analyzed (Participants) | 0

6. Primary Outcome: DTG PK Parameter Area Under the Concentration Time Curve (AUC0-24) Calculated Based on Intensive PK Samples Obtained From Individual Participants Enrolled in Arm 2 by Visit Day
Description: This evaluates the effect of RPT on the DTG PK parameter AUC 0-24h obtained from participants enrolled in Arm 2 at day 0 (DTG QD) and day 28 (DTG QD with 1HP). AUC 0-24h defines area under the concentration-time curve over the period of 24 hours post-dose estimated based on the fitted model.
Time Frame: Intensive DTG PK samples at pre-dose, 1h, 2h, 4h, 8h, 12h, 23h and 24h post-dose at days 0 and 28
Population: It was decided to not move forward with Arm 2 of the study and no participants were enrolled in Arm 2.
Arm/Group | Arm 2: DTG + INH + RPT
Number analyzed (Participants) | 0

7. Primary Outcome: DTG PK Parameter Minimum Plasma Concentration (Cmin) Determined Based on DTG Levels From Individual Participants in Arm 2 by Visit Day
Description: This evaluates the effect of RPT on the DTG PK parameter Cmin obtained from participants enrolled in Arm 2 at day 0 (DTG QD) and day 28 (DTG QD with 1HP). Cmin defines the model-predicted minimum concentration observed over the 24- hour DTG dosing interval.
Time Frame: Intensive DTG PK samples at pre-dose, 1h, 2h, 4h, 8h, 12h, 23h and 24h post-dose at days 0 and 28
Population: It was decided to not move forward with Arm 2 of the study and no participants were enrolled in Arm 2.
Arm/Group | Arm 2: DTG + INH + RPT
Number analyzed (Participants) | 0

8. Primary Outcome: DTG PK Parameter Ctrough Determined Based on DTG Levels From Individual Participants in Arm 2 at Day 28
Description: This evaluates the effect of RPT on the DTG PK parameter Ctrough obtained from participants enrolled in Arm 2 at day 28 (DTG QD with 1HP). Ctrough defines the observed non-model based minimum concentration observed over the 24- hour DTG dosing interval.
Time Frame: Intensive DTG PK samples at pre-dose, 1h, 2h, 4h, 8h, 12h, 23h and 24h post-dose at days 0 and 28
Population: It was decided to not move forward with Arm 2 of the study and no participants were enrolled in Arm 2.
Arm/Group | Arm 2: DTG + INH + RPT
Number analyzed (Participants) | 0

9. Secondary Outcome: Percentage of Participants in Arm 1 With an Occurrence of Grade 2 or Higher Adverse Event
Description: Arm 1 participants with an occurrence of an adverse event (laboratory value, sign/symptom, diagnosis) of grade 2 or higher on a scale of 1 to 5 where 5 is the most severe. Severity graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017. Participants were counted once at the highest grade.
Time Frame: From initiation of study treatment to day 28
Population: Participants who took at least one dose of RPT, at least one dose of INH, and at least 2 doses of DTG.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: DTG + INH + RPT
Number analyzed (Participants) | 36
Percentage of participants
  Grade 2 Adverse Event | 36 [21 to 54]
  Grade 3 Adverse Event | 6 [1 to 19]

10. Secondary Outcome: Percentage of Participants in Arm 1 Who Completed the Study
Description: Percentage of participants in Arm 1 who completed the study
Time Frame: From initiation of study to day 28
Population: Participants who took at least one dose of RPT, at least one dose of INH, and at least 2 doses of DTG.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: DTG + INH + RPT
Number analyzed (Participants) | 36
Percentage of participants | 89 [74 to 97]

11. Secondary Outcome: Percentage of Participants in Arm 1 Who Completed Study Drug Treatment
Description: Percentage of participants in Arm 1 who completed study drug treatment (DTG+1HP)
Time Frame: From initiation of study treatment to day 28
Population: Participants who took at least one dose of RPT, at least one dose of INH, and at least 2 doses of DTG.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1: DTG + INH + RPT
Number analyzed (Participants) | 36
Percentage of participants | 92 [78 to 98]

12. Secondary Outcome: Percentage of Participants in Arm 1 With HIV-1 RNA Levels >50 Copies/mL
Description: This evaluates the short-term impact on virologic suppression of DTG based ART when coadministered with 1HP by measuring the percentage of participants with plasma HIV-1 RNA levels >50 copies/mL at study day 28 (after 4 weeks of DTG+1HP) and study day 42 (14 days after completing study treatment).
Time Frame: Measured at Days 28 and 42
Population: All participants in who took at least one dose of study drugs and who had HIV-1 RNA data available.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: DTG + INH + RPT
Number analyzed (Participants) | 33
percentage of participants
  Percentage with HIV-1 RNA >50 copies/mL at day 28 | 3
  Percentage with HIV-1 RNA >50 copies/mL at day 42: number analyzed (Participants) | 32
  Percentage with HIV-1 RNA >50 copies/mL at day 42 | 0

13. Secondary Outcome: Percentage of Participants in Arm 2 With an Occurrence of Grade 2 or Higher Adverse Event
Description: Arm 2 participants with an occurrence of an adverse event (laboratory value, sign/symptom, diagnosis) of grade 2 or higher on a scale of 1 to 5 where 5 is the most severe. Severity graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017. Participants will be counted once at the highest grade.
Time Frame: From initiation of study treatment to day 28
Population: It was decided to not move forward with Arm 2 of the study and no participants were enrolled in Arm 2.
Arm/Group | Arm 2: DTG + INH + RPT
Number analyzed (Participants) | 0

14. Secondary Outcome: Percentage of Participants in Arm 2 Who Completed the Study
Description: Percentage of participants in Arm 2 who completed the study.
Time Frame: From initiation of study to day 28
Population: It was decided to not move forward with Arm2 of the study and no participants were enrolled in Arm 2.
Arm/Group | Arm 2: DTG + INH + RPT
Number analyzed (Participants) | 0

15. Secondary Outcome: Percentage of Participants in Arm 2 Who Completed Study Drug Treatment
Description: Percentage of participants in Arm 2 who completed study drug treatment (DTG+1HP).
Time Frame: From initiation of study treatment to day 28
Population: It was decided to not move forward with Arm2 of the study and no participants were enrolled in Arm 2.
Arm/Group | Arm 2: DTG + INH + RPT
Number analyzed (Participants) | 0

16. Secondary Outcome: Percentage of Participants in Arm 2 With HIV-1 RNA Levels >50 Copies/mL
Description: as for outcome 12
Time Frame: Measured at Days 28 and 42
Population: It was decided to not move forward with Arm2 of the study and no participants were enrolled in Arm 2.
Arm/Group | Arm 2: DTG + INH + RPT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From start of study treatment to study completion at Day 49 or premature study discontinuation.
Description: All participants who took at least one dose of RPT, at least one dose of INH, and at least 2 doses of DTG were included.
Arm/Group | Arm 1: DTG + INH + RPT
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 15/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: DTG + INH + RPT (N=36)
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 3
Conjunctivitis allergic (Eye disorders) | 1
Pyrexia (General disorders) | 1
COVID-19 (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 3
Glomerular filtration rate decreased (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT04272242/Prot_ICF_002.pdf
  • Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT04272242/SAP_001.pdf